CLINICAL TRIAL: NCT06332820
Title: In Patients With Obstructive Airway Disease, Investigate the Effects of Different Breathing Strategies and Pedaling Rates on the Physiological Response to Bicycle Exercise
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202401226RINB
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Airway Disease
Keywords: Obstructive airway disease; Cardiopulmonary exercise test
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The definition of obstructive airway disease is a ratio of the forced expiratory volume in one second (FEV1) to the forced vital capacity (FVC) of less than 0.7, which includes conditions such as chronic obstructive pulmonary disease, asthma, lymphangioleiomyomatosis, and bronchiolitis obliterans syndrome. For example, lung obstruction adversely affects many aspects of a patient's health, such as lung function and exercise capacity. Pulmonary rehabilitation is widely used in patients with obstructive airway disease, and the prescription of pulmonary rehabilitation depends on exercise capacity parameters such as peak oxygen uptake (peak VO2), peak workload, and anaerobic threshold. However, patients often have difficulty achieving training goals due to severe dyspnea during exercise. Dynamic hyperinflation is a common cause of dyspnea during exercise in patients with obstructive airway disease. Investigators aim to alleviate breathlessness by reducing dynamic hyperinflation, making it easier to achieve training goals. Methods to reduce dynamic hyperinflation include pursed lip breathing, reducing breathing rate to prolong expiratory time, using bronchodilators, and undergoing lung volume reduction surgery. Among these methods, reducing breathing rate to prolong expiratory time may be the most feasible, and investigators aim to change the rhythm and pace of breathing by adjusting the pedal rate of cycling exercise. The pedaling rate is typically set at 60 revolutions per minute. The European Respiratory Society recommended a pedal rate range of 40-70 revolutions per minute in 2019. There is still no consensus on the relationship between pedal rate and respiratory rate. This prospective observational study, using a crossover design, aims to investigate the effects of pedal rate during exercise testing on dynamic hyperinflation and exercise capacity in patients with obstructive airway disease.

DETAILED DESCRIPTION:
Obstructive airway disease is defined as forced expiratory volume in one second (FEV1) / forced vital capacity (FVC) <0.7. It includes chronic obstructive pulmonary disease (COPD), asthma, lymphangioleiomyomatosis (LAM) and bronchiolitis obliterans syndrome. Pulmonary rehabilitation is widely utilized in patients with obstructive airway disease. Comprehensive intervention based on a thorough patient assessment followed by patient-tailored therapies that include, but are not limited to, exercise training, education, and behavior change, designed to improve the physical and psychological condition of people. The exercise prescription for pulmonary rehabilitation is often determined based on exercise capacity. The exercise capacity includes peaked VO2 (oxygen consumption), peaked work rate, and anaerobic threshold. They are all measured in cardiopulmonary exercise test (CPET). However, patients often struggle to achieve training goals due to severe dyspnea. Dynamic hyperinflation is a common cause of shortness of breath on exertion in obstructive airway disease.

Generally, end-expiratory lung volume (EELV) is relative constant during exercise. Inspiratory capacity (IC) is increasing during exercise. The IC maneuver is used to monitor exercise-induced dynamic hyperinflation. Dynamic hyperinflation caused by air trapping, which increases residual air volume, is a common cause of shortness of breath on exertion in obstructive lung disease. There are many diagnostic criteria, including a decrease in dynamic IC of >140mL, a decrease of ≥5% in IC during maximal exercise, or a decrease of ≥10% in IC during maximal exercise. In a prospective observational study, dynamic hyperinflation occurred at a higher prevalence (55%) in patients with LAM. Dynamic hyperinflation was associated with a reduction in FEV1 and higher dyspnea intensity at exercise cessation (R = -0.53, P-value < 0.001). COPD patients develop dynamic hyperinflation during symptom-limited incremental work exercise with cycle ergometer. The increase in EELV seems to be the best predictor of dyspnea.

The pedaling rate is typically set at 60 revolutions per minute in National Taiwan University Hospital. The average respiratory rate for a total of 31 patients is 29 breaths per minute. 2019 European respiratory society suggested that maintaining over a wide range of pedaling rates (40-70 revolutions per minute) in CPET. The evidence of the optimal pedaling rate during exercise obstructive airway disease is limited. The current consensus remains inconclusive on whether a lower pedaling rate will result in a reduction of breathing speed, subsequently improving dynamic hyperinflation, and ultimately leading to an improvement in exercise capacity. This prospective observational study, employing a crossover design, aims to investigate the impact of pedaling rate during exercise tests on dynamic hyperinflation and exercise capacity in individuals with obstructive airway disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18

Exclusion Criteria:

* Coronary angiography via femoral artery in recent 3 days
* Central venous catheter in femoral vein
* The patient couldn't walk over 20 meters
* Lower limb arthropathy
* Unclear consciousness and the patient couldn't cooperate well
* SPO2 < 85%
* Acute coronary syndrome in recent 1 month
* Respiratory failure or unstable hemodynamics
* Pneumothorax or bronchial fistula
* Acute exacerbation in recent 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obstructive airway disease patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Inspiratory capacity during exercise | During the cardiopulmonary exercise test
  Inspiratory capacity during exercise

SECONDARY OUTCOMES:
Change of FEV1 and symptoms | During the cardiopulmonary exercise test
  Change of FEV1 and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Yu Liao, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No